CLINICAL TRIAL: NCT01400217
Title: HFA Beclomethasone in Asthma, a General Practice Research Database Study: Real-life Observational Evaluation of Extra-fine With Standard Particle Size Beclometasone Dipropionate Using the Propellant Hydrofluoroalkane 134a for the Management of Asthma in a Representative UK Primary Care Population
Brief Title: Qvar Versus Clenil, a General Practice Research Database Study
Status: Completed | Type: Observational
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Principal Investigator, David Price, Professor David Price, Research in Real-Life Ltd
Other Study IDs: 007/11
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Asthma
Keywords: Primary Care; Particle size; beclomethasone dipropionate; Asthma Management; Maintenance Therapy; Metered-Dose Inhaler
MeSH Terms: conditions — Asthma | interventions — Beclomethasone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- IPDI EF HFA-BDP: Patients initiating inhaled corticosteroid therapy as extra-fine HFA-BDP MDI at the index date
  Interventions: Drug: extra fine particle hydrofluoroalkane beclomethasone dipropionate via metered dose inhaler
- IPDI SP HFA-BDP: Patients initiating inhaled corticosteroid therapy as standard particle HFA-BDP MDI at the index date
  Interventions: Drug: standard particle particle hydrofluoroalkane beclomethasone dipropionate via metered dose inhaler
- IPDA SP HFA-BDP: Patients increased inhaled corticosteroid therapy as standard particle HFA-BDP MDI at the index date
  Interventions: Drug: standard particle particle hydrofluoroalkane beclomethasone dipropionate via metered dose inhaler
- IPDA EF HFA-BDP: Patients increased inhaled corticosteroid therapy as extra fine particle HFA-BDP MDI at the index date
  Interventions: Drug: extra fine particle hydrofluoroalkane beclomethasone dipropionate via metered dose inhaler
- IPDS SP HFA-BDP: Patients increased inhaled corticosteroid therapy as standard particle HFA-BDP MDI at the index date
  Interventions: Drug: standard particle particle hydrofluoroalkane beclomethasone dipropionate via metered dose inhaler
- IPDS EF HFA-BDP: Patients increased inhaled corticosteroid therapy as extrafine particle HFA-BDP MDI at the index date
  Interventions: Drug: extra fine particle hydrofluoroalkane beclomethasone dipropionate via metered dose inhaler

INTERVENTIONS:
Drug: extra fine particle hydrofluoroalkane beclomethasone dipropionate via metered dose inhaler — IPDI cohort intervention = initiation of intervention drug; IPDS cohort intervention = switching from baseline inhaled corticosteroid therapy to intervention drug without a change in baseline inhaled corticosteroid dose; IPDA cohort intervention = increase in baseline inhaled corticosteroid drug as intervention drug
  Other Names: Qvar
  Groups: IPDA EF HFA-BDP; IPDI EF HFA-BDP; IPDS EF HFA-BDP
Drug: standard particle particle hydrofluoroalkane beclomethasone dipropionate via metered dose inhaler — IPDI cohort intervention = initiation of intervention drug; IPDS cohort intervention = switching from baseline inhaled corticosteroid therapy to intervention drug without a change in baseline inhaled corticosteroid dose; IPDA cohort intervention = increase in baseline inhaled corticosteroid drug as intervention drug
  Other Names: Fostair
  Groups: IPDA SP HFA-BDP; IPDI SP HFA-BDP; IPDS SP HFA-BDP

SUMMARY:
This study will compare the absolute and relative effectiveness of asthma management in patients on inhaled corticosteroid (ICS) maintenance therapy as either extra-fine-particle or larger-particle formulation beclomethasone dipropionate (BDP) via metered-dose inhalers (MDIs) using the propellant hydrofluoroalkane propellant (HFA-BDP), namely Qvar® MDI compared with Clenil® MDI.

DETAILED DESCRIPTION:
Current asthma guidelines in the UK are underpinned by evidence derived from randomised controlled trials (RCTs). Although RCT data are considered the gold standard, patients recruited to asthma RCTs are estimated to represent less than 10% of the UK's asthma population. The poor representation of the asthma population is due to a number of factors, such as tightly-controlled inclusion criteria for RCTs. There is, therefore, a need for more representative RCTs and real-life observational studies to inform existing guidelines and help optimise asthma outcomes.

In response to the Montreal Protocol's ruling to phase out ozone-depleting chlorofluorocarbon (CFC) propellants in asthma inhalers, several hydrofluoroalkane-134a-propellant (HFA-) formulations of BDP have been developed. Two branded generic formulations currently available in the UK are Qvar® (Teva Pharmaceutical Industries Ltd) - an extra-fine-particle (~1.1 microns) HFA-BDP (solution) formulation and Clenil® (Chiesi Limited) - a larger particle (~2.9 microns) HFA-BDP (suspension) formulation.

The extra-fine particle formulation HFA-BDP formulation (Qvar®) has been shown to improve total and small airway deposition relative to CFC-BDP. As a result of the more even distribution through both the large and small airways of the lungs and data from short-term randomised clinical trials (RCTs), Qvar® dosing is recommended at approximately one half the dose of traditional CFC-BDP (average particle size ~3.5 microns). However, the larger-particle Clenil® is recommended for prescribing at the same dose as traditional CFC-BDP.

Further studies are required to understand whether the differences in particle size and airway distribution have an impact on asthma outcomes over the long-term.

This observational study will investigate the real-world effectiveness of extra-fine HFA-BDP (Qvar®) as compared with larger-particle HFA-BDP (Clenil®) in patients with asthma who: were new to ICS therapy; received an increase in their ICS dose, or switched / changed baseline ICS therapy to HFA-BDP with no change in BDP-equivalent ICS dose. We hypothesise that differences in effectiveness might become apparent over the longer term through a retrospective database analysis of one-year outcomes for the diverse patient population seen in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Aged: 4-80 years
* Paediatric cohort (aged 4-11 years), and
* Adult cohort (aged 12-80 years )
* Evidence of asthma and current asthma therapy:
* All cohorts (IPDI, IPDS, IPDA):

  * a diagnostic code for asthma, and / or *≥2 prescriptions for asthma at different points in time during the prior year and/or IPDI only: ≥2 prescriptions for asthma therapies during the outcome year, including ≥1 ICS prescription in addition to that received at IPD

IPDA and IPDS only:

* 1 ICS prescription in the baseline year, and
* 1 other asthma prescription during the baseline year.

  *Evidence of "current therapy":
* 2 prescription for ICS during the outcome year (i.e. ≥1 prescription in addition to the prescription at index date

  * Have at least one year of up-to-standard (UTS) baseline data (prior to the IPD) and at least one year of UTS outcome data (following the IPD).

Exclusion Criteria:

* Had a COPD read code at any time; and/or
* Had any chronic respiratory disease, except asthma, at any time; and/or
* Patients on maintenance oral steroids during baseline year
* Received a combination inhaler in addition to a separate ICS inhaler in the baseline year; and/or
* Received ICS therapy during baseline year via DPI (IPDA and IPDS cohorts only).
* If they received multiple ICS prescriptions on the same day at IPD or immediately before

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients are aged between 4-80 years and have evidence of asthma and subsequent therapy.
Sampling Method: Non-Probability Sample
Enrollment: 56985 (Actual)
Dates: Start 1991-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Severe asthma exacerbation (ATS/ERS based defn) | 1 year
  Exacerbation defined as:
  (i) Respiratory-related:
  1. Hospital attendance / admissions OR
  2. A&E attendance OR (ii) Use of acute oral steroids**
Primary composite asthma control | 1 year
  Where control is defined as absence of:
  (i) Respiratory-related:
  1. Hospital attendance or admission
  2. A&E attendance, OR
  3. Out of hours attendance, OR
  4. Out-patient department attendance (ii) GP consultations for lower respiratory tract infection (iii) Prescriptions for acute courses of oral steroids

SECONDARY OUTCOMES:
Exacerbation definition based on clinical experience | 1 year
  Defined as:
  (i) Respiratory-related:
  1. Hospital attendance / admissions OR
  2. A&E attendance OR
  3. Out of hours consultation OR
  4. GP consultation OR (ii) Use of acute oral steroids
Asthma control + SABA usage | 1 year
  Where control requires the absence of:
  (i) Respiratory-related:
  1. Hospital attendance or admission
  2. A&E attendance, OR
  3. Out of hours consultation, OR
  4. Out-patient department attendance (ii) GP consultations for lower respiratory tract infection (iii) Prescriptions for acute courses of oral steroids (iv) Average daily prescribed dose of ≤200mcg salubtamol / ≤500mcg terbutaline
Treatment success | 1 year
  (i) Control
  a. No respiratory-related: i. Hospital attendance or admission ii. A&E attendance, OR iii. Out of hours consultation, OR iv. Out-patient department attendance b. No GP consultations for lower respiratory tract infection (ii) No prescriptions for acute courses of oral steroids (iii) No additional or change in therapy
  1. Increased dose of ICS (≥50% increase), and/or
  2. Change in ICS and/or
  3. Change in delivery device, and/or
  4. Use of additional therapy as defined by: LABA, theophylline, leukotreine receptor antagonists (LTRAs).
Asthma-related hospitalisations | 1 year
  Defined as sum of:
  (i) Definite: Hospitalisations coded with an asthma read code (ii) Definite + Probable: Hospitalisations with an asthma read code + uncoded hospitalisations occurring within a 7-day window (either side of the hospitalisation date) of an asthma read code
Respiratory hospitalisations | 1 year
  Defined as the sum of:
  (i) Definite: Hospitalisations coded with a lower respiratory code (ii) Definite + Probable: Hospitalisations with an asthma read code + uncoded hospitalisations occurring within a 7-day window (either side of the hospitalisation date) of a lower respiratory read code
SABA usage | 1 year
  Average daily dosage during outcome year - outcome SABA usage will be categorised within ranges used to match baseline SABA use to optimise matching of the treatment arms.
ICS compliance | 1 year
  Based on prescription refills
Oral Thrush | 1 year
  Defined as:
  (i) Topical oral anti-fungal prescriptions, and / or (ii) Coded for oral candidiasis

CONTACTS AND LOCATIONS:
Overall Officials: David Price, MD, Principal Investigator — Company Director
Locations (1):
- Research in Real Life Ltd, Cawston, Norfolk, United Kingdom

REFERENCES:
- [Background] Herland K, Akselsen JP, Skjonsberg OH, Bjermer L. How representative are clinical study patients with asthma or COPD for a larger "real life" population of patients with obstructive lung disease? Respir Med. 2005 Jan;99(1):11-9. doi: 10.1016/j.rmed.2004.03.026. PMID 15672843
- [Background] Travers J, Marsh S, Caldwell B, Williams M, Aldington S, Weatherall M, Shirtcliffe P, Beasley R. External validity of randomized controlled trials in COPD. Respir Med. 2007 Jun;101(6):1313-20. doi: 10.1016/j.rmed.2006.10.011. Epub 2006 Nov 17. PMID 17113277
- [Background] Appleton SL, Adams RJ, Wilson DH, Taylor AW, Ruffin RE; North West Adelaide Cohort Health Study Team. Spirometric criteria for asthma: adding further evidence to the debate. J Allergy Clin Immunol. 2005 Nov;116(5):976-82. doi: 10.1016/j.jaci.2005.08.034. PMID 16275363
- [Background] Vanden Burgt JA, Busse WW, Martin RJ, Szefler SJ, Donnell D. Efficacy and safety overview of a new inhaled corticosteroid, QVAR (hydrofluoroalkane-beclomethasone extrafine inhalation aerosol), in asthma. J Allergy Clin Immunol. 2000 Dec;106(6):1209-26. doi: 10.1067/mai.2000.111582. PMID 11112914
- [Background] Leach CL, Davidson PJ, Hasselquist BE, Boudreau RJ. Influence of particle size and patient dosing technique on lung deposition of HFA-beclomethasone from a metered dose inhaler. J Aerosol Med. 2005 Winter;18(4):379-85. doi: 10.1089/jam.2005.18.379. PMID 16379614
- [Background] Leach CL, Davidson PJ, Boudreau RJ. Improved airway targeting with the CFC-free HFA-beclomethasone metered-dose inhaler compared with CFC-beclomethasone. Eur Respir J. 1998 Dec;12(6):1346-53. doi: 10.1183/09031936.98.12061346. PMID 9877489
- [Background] Busse WW, Brazinsky S, Jacobson K, Stricker W, Schmitt K, Vanden Burgt J, Donnell D, Hannon S, Colice GL. Efficacy response of inhaled beclomethasone dipropionate in asthma is proportional to dose and is improved by formulation with a new propellant. J Allergy Clin Immunol. 1999 Dec;104(6):1215-22. doi: 10.1016/s0091-6749(99)70016-3. PMID 10589004
- [Background] Davies RJ, Stampone P, O'Connor BJ. Hydrofluoroalkane-134a beclomethasone dipropionate extrafine aerosol provides equivalent asthma control to chlorofluorocarbon beclomethasone dipropionate at approximately half the total daily dose. Respir Med. 1998 Jun;92 Suppl A:23-31. doi: 10.1016/s0954-6111(98)90214-1. PMID 9850360
- [Background] Gross G, Thompson PJ, Chervinsky P, Vanden Burgt J. Hydrofluoroalkane-134a beclomethasone dipropionate, 400 microg, is as effective as chlorofluorocarbon beclomethasone dipropionate, 800 microg, for the treatment of moderate asthma. Chest. 1999 Feb;115(2):343-51. doi: 10.1378/chest.115.2.343. PMID 10027430
- [Background] IBM SPSS Statistics. 2010. Statistics family. Available online at: www.spss.com/uk/software/statistics/
- [Background] AS Institute Inc. 2010. Statistical Analysis with SAS/STAT Software. Available online at: www.SAS.com/offices/europe/uk/technologies/analytics/statistics/stat/ondex.html
- [Derived] Price D, Thomas M, Haughney J, Lewis RA, Burden A, von Ziegenweidt J, Chisholm A, Hillyer EV, Corrigan CJ. Real-life comparison of beclometasone dipropionate as an extrafine- or larger-particle formulation for asthma. Respir Med. 2013 Jul;107(7):987-1000. doi: 10.1016/j.rmed.2013.03.009. Epub 2013 May 3. PMID 23643486